CLINICAL TRIAL: NCT04423523
Title: Plasma Levels of Danger-Associated Molecular Patterns (DAMPs) in Young Children After Cardiac Surgery Under Cardiopulmonary Bypass (IMMUNOPED 2)
Brief Title: Plasma Levels of Danger-Associated Molecular Patterns in Young Children After Cardiac Surgery Under Cardiopulmonary Bypass
Acronym: IMMUNOPED2
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC19_0402
Record Dates: First submitted 2020-05-14; First posted 2020-06-09 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2024-12

CONDITIONS: Cardiac Surgical Procedure
Keywords: cardiopulmonary bypass; immunosuppression; infant; immunosuppression; infant

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study population: The study population must correspond to the research inclusion criteria: Patient admitted to pediatric intensive care at Nantes University Hospital after cardiac surgery on bypass grafts
  Interventions: Diagnostic Test: Blood drop sampling

INTERVENTIONS:
Diagnostic Test: Blood drop sampling — For each patient included, 1 additional EDTA blood tube (2 ml) will be collected for research purposes at different times (4 visits), and 1 PAXgene-type tube adapted for pediatric collection of only 500 μl (2 visits).

SUMMARY:
The investigators have previously reported that cardiac surgery with CPB ( cardiopulmonary bypass) in young infants induced a drastic reduction in mHLA-DR ( Human Leucocyte Antigen) expression, which represents one of innate immune mediator. Danger-Associated Molecular Patterns (DAMPs) can elicit immune response and may subsequentely induce an immune-suppressed state. The investigators hypothesize that CPB causes excessive DAMP release, leading to the development of immune suppression. Thus, DAMPs release will be assessed in patients undergoing CBP, and consequences on immune suppression will be evaluated.

DETAILED DESCRIPTION:
Plasma levels of heat shock protein (HSP 70), high mobility group box (HMGB1), S100A9 and IL-33 will be measured at four time points (prior to the onset of CPB, Hour 6 postoperative, day 1 and day 3 after surgery). HLA-DR gene expression will be determined before surgery and at day 3 postoperative. The direct effect of DAMPs release and immune suppression will be assessed by in vitro experiments.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted to pediatric intensive care at Nantes University Hospital after cardiac surgery with bypass graft
* Age ≤ 3 months corrected age. Control group: patients less than 3 months old following cardiac surgery without CEC or digestive surgery with a central venous catheter.

Exclusion Criteria:

* Futility of care with cessation of blood tests as part of a limitation of active therapies;
* Absence of parents for information
* Refusal of parents after information (Lack of parental consent)
* Blood volume collected for medical purposes incompatible with the needs of the research

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All patients admitted to pediatric resuscitation at the Nantes University Hospital after cardiac surgery under CEC ( extra-corporal circulation) and aged less than 3 months meeting the criteria for inclusion and non-inclusion of the study will be included. We can objectify the recruitment of 80 patients in total over 3 years.
  Since natural evolution (variation of rates and their kinetics) of the secretion of different DAMPs during the first months of life is unknown, the investigators added a control group to know the expression and kinetics of DAMPs outside cardiac surgery under CEC. This control group will be defined by infants under 3 months of age undergoing heavy digestive surgery and having a central venous catheter to facilitate access to blood samples (n = 20).
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2025-12-02 (Actual)

PRIMARY OUTCOMES:
Plasma levels of heat shock protein (HSP 70), high mobility group box (HMGB1), S100A9 and IL-33 before and after CBP. | prior to the onset of CPB, 6 hours, day 1 and day 3 after surgery
  Change of plasma levels of DAMPs after cardiopulmonary bypass Plasma levels of heat shock protein (HSP 70), high mobility group box (HMGB1), S100A9 and IL-33 before and after CBP.

SECONDARY OUTCOMES:
Effect of DAMPs on immune function:In vitro change of HLA-DR expression. | 6 hours after surgery
  In vitro change of HLA-DR expression induced by plasma containing different concentrations of DAMPs.
Effect of DAMPs on immune function:Secretion of IL-10 ( Interleukine 10). | 6 hours after surgery
  Secretion of IL-10 by different immune cells induced by plasma containing different concentrations of DAMPs.

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Chenouard, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France